CLINICAL TRIAL: NCT04790396
Title: Carotid Ultrasound Under Pulsed-wave Doppler Mode to Check the Pulse in Cardiopulmonary Arrest Patients.
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202010082RINB
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient presenting at emergent department with cardiac arrest
  Interventions: Device: Carotid ultrasound under pulsed-wave doppler mode

INTERVENTIONS:
Device: Carotid ultrasound under pulsed-wave doppler mode — Carotid ultrasound under pulsed-wave doppler mode to check whether carotid pulse is present

SUMMARY:
It's crucial to determine whether a pulse is present or not in patient with cardiac arrest. But more and more studies have shown that manual palpation is unreliable for detecting pulse 1-4. Failure to detect pulselessness may cause delay of chest compression and directly affect the patient's outcome. Likewise, failure to rapidly detect return of spontaneous circulation may cause prolonged chest compression and increase associated injury during resuscitation.

More and more studies have demonstrated that echo guided pulse detection is feasible 5-7. The aim of our study is to check carotid pulse via ultrasound. This is a prospective study and the patient selection is in-hospital or out of hospital cardiac arrest. A curvilinear ultrasonography transducer is used and placed transversely on either right/left carotid artery under pulsed-wave doppler mode to check whether the pulse is present or not. The result of ultrasonography will be compared with manual palpation and to determine the accuracy and effectiveness of clinical usage.

ELIGIBILITY:
Inclusion Criteria:

* any patient presenting at ER with cardiac arrest older than 20 years-old

Exclusion Criteria:

* younger than 20 years-old
* patient who is pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any patient presenting at ER with cardiac arrest older than 20 years-old, including trauma or non-trauma cardiac arrest, in-hospital or out-of-hospital cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Carotid ultrasound under pulsed-wave doppler compared with manual palpation | 5 seconds during pulse check period of resuscitation
  The result of ultrasonography will be compared with manual palpation and to determine the accuracy（e.g., no pulse under manual palpation but positive pulse-wave finding）of clinical usage.
Carotid ultrasound under pulsed-wave doppler compared with manual palpation | 5 seconds during pulse check period of resuscitation
  The result of ultrasonography will be compared with manual palpation and to determine the effectiveness (e.g., the time need to confirm whether pulse is present or not under manual palpation and ultrasound) of clinical usage.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bahr J, Klingler H, Panzer W, Rode H, Kettler D. Skills of lay people in checking the carotid pulse. Resuscitation. 1997 Aug;35(1):23-6. doi: 10.1016/s0300-9572(96)01092-1. PMID 9259056
- [Result] Eberle B, Dick WF, Schneider T, Wisser G, Doetsch S, Tzanova I. Checking the carotid pulse check: diagnostic accuracy of first responders in patients with and without a pulse. Resuscitation. 1996 Dec;33(2):107-16. doi: 10.1016/s0300-9572(96)01016-7. PMID 9025126
- [Result] Moule P. Checking the carotid pulse: diagnostic accuracy in students of the healthcare professions. Resuscitation. 2000 May;44(3):195-201. doi: 10.1016/s0300-9572(00)00139-8. PMID 10825620
- [Result] Liberman M, Lavoie A, Mulder D, Sampalis J. Cardiopulmonary resuscitation: errors made by pre-hospital emergency medical personnel. Resuscitation. 1999 Sep;42(1):47-55. doi: 10.1016/s0300-9572(99)00082-9. PMID 10524730
- [Result] Badra K, Coutin A, Simard R, Pinto R, Lee JS, Chenkin J. The POCUS pulse check: A randomized controlled crossover study comparing pulse detection by palpation versus by point-of-care ultrasound. Resuscitation. 2019 Jun;139:17-23. doi: 10.1016/j.resuscitation.2019.03.009. Epub 2019 Mar 20. PMID 30902687
- [Result] Simard RD, Unger AG, Betz M, Wu A, Chenkin J. The POCUS Pulse Check: A Case Series on a Novel Method for Determining the Presence of a Pulse Using Point-of-Care Ultrasound. J Emerg Med. 2019 Jun;56(6):674-679. doi: 10.1016/j.jemermed.2019.02.013. Epub 2019 Apr 16. PMID 31003817
- [Result] Germanoska B, Coady M, Ng S, Fermanis G, Miller M. The reliability of carotid ultrasound in determining the return of pulsatile flow: A pilot study. Ultrasound. 2018 May;26(2):118-126. doi: 10.1177/1742271X17753467. Epub 2018 Jan 29. PMID 30013612